CLINICAL TRIAL: NCT03711643
Title: Hypnosis Mask: a New Approach to Management of Pain in Medical Imaging
Acronym: HYPNOTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017_84; 2018-A01673-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2023-02

CONDITIONS: Prostatic Diseases
Keywords: prostatic biopsies echo-guided; Pain measurement; Anxiety assessment
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimizing pain management (Experimental): An experimental group receive a standard pain management and benefit the hypnotic mask (Hypnos pro).
  Interventions: Procedure: Periprostatic nerve block; Device: hypnosis mask
- standard pain management (Active Comparator)
  Interventions: Procedure: Periprostatic nerve block

INTERVENTIONS:
Procedure: Periprostatic nerve block — 4 injections of 2 cc of lidocaine for a Periprostatic nerve block
Device: hypnosis mask — The mask HYPNOS pro stimulates the imagination of the user by means of 6 diodes among 3 by eye.
  Just before the introduction of ultrasound probe, the patient put the hypnotic mask and choose a session.Twenty minutes after the removal of the probe, an healthworker assess the painful patient with the visual analogue scale VAS, after this the patient fulfill the STATE- TRAIT Anxiety Inventory (STAI) form Y-A.
  Arms: Optimizing pain management

SUMMARY:
The prostatic biopsies echo-guided are a painful and stressful. The purpose is to test a new medical device created recently, " Hypnos-Pro ", wich uses connected technologies. This connected device is a mask with diodes coupled with an audio headset and a touch pad. This connected mask is an another option to induce an hypnotic state for our patients. the objective is to value hypnotic mask effectiveness, to reduce the level pain and anxiety for the patients who benefit a prostatic biopsies echo-guided with local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for prostate biopsies
* Having accepted and signed the consent, for performing a prostate biopsy ultrasound examination
* No contraindication to the gesture
* Supporting the left lateral decubitus

Exclusion Criteria:

* Patient isolation contact / droplets
* Patient with hearing and / or epilepticus and / or dementia and / or having a history of stroke and / or allergic to lidocaine
* Person unable to consent, or benefiting from a system of legal protection (tutelage / curatorship).
* Patients with epileptic seizures.
* Patients with known allergies to plastics and other resins that may develop allergic contact dermatitis.
* Patients who are hypersensitive to radio frequency.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Visual analogic Scale | at 20 minutes after the removal of the probe
  Measure the pain in the scale from 0 to 10

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory ou STAI forme Y-A | Baseline, at 20 minutes after the removal of the probe
Percentage of positive response of satisfaction of the patient | at 20 minutes after the removal of the probe
  The question is: Would you do prostate biopsy punctures under the same conditions in a month? (Yes: effective method, No: ineffective method).
Percentage of positive response of satisfaction of the operator | at 20 minutes after the removal of the probe
  The question is: In your opinion, has the gesture been made optimally? (Yes/ No).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Puech, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France